CLINICAL TRIAL: NCT00769418
Title: A Double-Blind, Randomized, Placebo-Controlled, Multi-Panel, Multiple Oral Dose Study, to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of MK0822 in Healthy Male and Postmenopausal Female Subjects
Brief Title: Study of Multiple Oral Doses of Odanacatib (MK0822) in Healthy Adults (0822-002)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0822-002; MK0822-002; 2008_558
Record Dates: First submitted 2008-10-06; First posted 2008-10-09 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — odanacatib

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): odanacatib (MK0822)
  Interventions: Drug: odanacatib
- 2 (Placebo Comparator): placebo to odanacatib (MK0822)
  Interventions: Drug: Comparator: Placebo

INTERVENTIONS:
Drug: odanacatib — Panels A, B, C, and D will enroll males only; Panels E, F, and G will enroll females only.
  Panel A: odanacatib tablets 2.5 mg qd for 14 days.
  Panel B: odanacatib tablets 5 mg qd for 14 days.
  Panel C: odanacatib tablets 10 mg qd for 14 days.
  Panel D: odanacatib tablets 25 mg qd for 14 days.
  Panel E: odanacatib tablets 0.5 mg qd for 21 days.
  Panel F: odanacatib tablets 2.5 mg qd for 21 days.
  Panel G: odanacatib tablets 10 mg qd for 21 days.
  Other Names: MK0822
  Arms: 1
Drug: Comparator: Placebo — Panels A, B, C, and D will enroll males only; Panels E, F, and G will enroll females only.
  Panel A: placebo to odanacatib tablets 2.5 mg qd for 14 days.
  Panel B: placebo to odanacatib tablets 5 mg qd for 14 days.
  Panel C: placebo to odanacatib tablets 10 mg qd for 14 days.
  Panel D: placebo to odanacatib tablets 25 mg qd for 14 days.
  Panel E: placebo to odanacatib tablets 0.5 mg qd for 21 days.
  Panel F: placebo to odanacatib tablets 2.5 mg qd for 21 days.
  Panel G: placebo to odanacatib tablets 10 mg qd for 21 days.
  Arms: 2

SUMMARY:
This study will assess the safety, tolerability, pharmacokinetics, and pharmacodynamics of once-daily multiple-dose administration of odanacatib (MK0822).

ELIGIBILITY:
Inclusion Criteria:

* Subject is a male between the ages of 18 and 45 or a female less than or equal to 70 years of age
* Females must be past menopause
* Subject is a nonsmoker
* Subject is willing to avoid excessive alcohol consumption during the study and is willing to avoid alcohol entirely for 24 hours prior to drug administration and during PK sampling
* Subject is willing to refrain from consuming grapefruit or grapefruit juice

Exclusion Criteria:

* Subject has a history of multiple/severe allergies to drugs or food
* Subject has donated blood within 4 weeks of starting the study
* Subject has a history of metabolic bone disease, urolithiasis, or bisphosphonate treatment
* Subject has any infections or any condition leading to immune problems, including HIV
* Subject regularly uses illegal drugs
* Subject consumes more than 3 alcoholic beverages per day
* Subject drinks 4 or more caffeinated beverages per day
* Subject uses any prescription or nonprescription medications

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2004-09; Primary Completion 2004-12 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of multiple oral doses of MK0822 | After 14 days of treatment for men and 21 days for women

SECONDARY OUTCOMES:
PK profile of MK0822 | predose and at selected time intervals postdose

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Stoch SA, Zajic S, Stone J, Miller DL, Van Dyck K, Gutierrez MJ, De Decker M, Liu L, Liu Q, Scott BB, Panebianco D, Jin B, Duong LT, Gottesdiener K, Wagner JA. Effect of the cathepsin K inhibitor odanacatib on bone resorption biomarkers in healthy postmenopausal women: two double-blind, randomized, placebo-controlled phase I studies. Clin Pharmacol Ther. 2009 Aug;86(2):175-82. doi: 10.1038/clpt.2009.60. Epub 2009 May 6. PMID 19421185